CLINICAL TRIAL: NCT05809401
Title: "Assessment and Treatment of Communicative Pragmatic Abilities in Neurological and Psychiatric Disorders: Feasibility and Clinical Efficacy (PATHS)"
Brief Title: Pragmatic Assessment and Treatment for the Health System
Acronym: PATHS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Camillo, Venezia, Italy (Other)
Collaborators: IRCCS San Raffaele (Other); Istituto Universitario di Studi Superiori Pavia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019.10
Record Dates: First submitted 2023-03-02; First posted 2023-04-12 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Stroke; Traumatic Brain Injury; Schizophrenia
MeSH Terms: conditions — Stroke; Brain Injuries, Traumatic; Schizophrenia | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRAGMACOM (Experimental): An experimental treatment for pragmatic disorders characterized by activities that focus on conversational rules and on understanding figurative language. The treatment is already tested on Schizophrenic patients.
  Interventions: Behavioral: Pragmatic Rehabilitation
- Standard Neuropsychological Treatment (Active Comparator): The standard treatment for neuropsychological disorders is administered to RHD, and TBI patients in the IRCCS San Camillo Hospital, which consists mostly of attentional training.
  Interventions: Behavioral: Neuropsychological Rehabilitation

INTERVENTIONS:
Behavioral: Pragmatic Rehabilitation — A series of behavioral activities to improve specific pragmatic abilities in patients
  Other Names: Pragmatic language Rehabilitation
  Arms: PRAGMACOM
Behavioral: Neuropsychological Rehabilitation — A series of behavioral activities to improve general aspect of cognition, with a specific focus on attentional abilities.
  Other Names: Cognitive Rehabilitation
  Arms: Standard Neuropsychological Treatment

SUMMARY:
The project goal is to promote a feasible and effective approach to communicative disorders in neurological and psychiatric populations, focused on the pragmatics of language. Pragmatics allows speakers to use and interpret language in context and to engage in successful communication. Pragmatic language disorder is widespread in clinical conditions and causes reduced social interactions and lower quality of life for both patients and their family. Yet it is seldom considered in assessment and rehabilitation.

DETAILED DESCRIPTION:
The project aims at developing a comprehensive approach for the assessment and treatment of pragmatic impairment in neurological disease. It consists of three Work Packages:

* The aim of WP1 is to develop a short test of pragmatic abilities. 200 healthy participants will be enrolled for this WP, and the same test will be administered to 40 patients with right hemisphere damage, 40 with traumatic brain injury, and 50 with Schizophrenia.
* The aim of WP2 is to test the efficacy of a novel treatment for pragmatic disorder. 32 patients will be enrolled (16 for each patient group) and allocated (via Randomized Control Trial) to a standard treatment or to a novel treatment for pragmatic disorders. Only RHD and TBI will take part to this WP.
* The aim of WP3 is to better clarify the neural correlates of pragmatic abilities. All patients will undergo an high density EEG recording session, and their brain activity will be correlated with performance on neuropsychological tests and on pragmatic impairment. The RHD and TBI patients enrolled for WP2 will undergo a session of hd-EEG also at the end of rehabilitation to monitor brain changes after treatment.

ELIGIBILITY:
Inclusion Criteria:

Healthy participants

* no neurological disorder
* written informed consent Right Hemisphere Damage (RHD)
* unilateral stroke
* first stroke
* no comorbidities with psychiatric disorders
* written informed consent TBI
* traumatic brain injury
* written informed consent

Schizophrenia:

* Diagnosis of Schizophrenia
* written informed consent

Exclusion Criteria:

* Important comorbidities that may affect results

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2019-11-13 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in APACS-Brief scores (Assessment of Pragmatic Abilities and Cognitive Substrates - Brief). | for healthy participants and all patients only t0 (immediatly after enrollment. For patients selected for WP2, T0 (after enrollment, as baseline) and T1 (after the treatment, that is after 1.5 months on average)
  A short test on pragmatic abilities. Scores range from 0 to 1. Higher values indicates better score

SECONDARY OUTCOMES:
Change in EEG (Electroencephalography) activity - ASSR (Auditory Steady State Response) | for healthy participants and all patients only t0 (immediatly after enrollment. For patients selected for WP2, T0 (after enrollment, as baseline) and T1 (after the treatment, that is after 1.5 months on average)
  EEG activity for ASSR is measured as power change in 40 Hz frequency as compared to baseline (time window from -100 to 0 ms). Score is unbounded. Higher values indicate better score (i.e., higher synchronization)
Change in EEG (Electroencephalography) activity - MMN (Mismatch Negativity) | for healthy participants and all patients only t0 (immediatly after enrollment. For patients selected for WP2, T0 (after enrollment, as baseline) and T1 (after the treatment, that is after 1.5 months on average)
  EEG activity for MMN is measured as average voltage deflection in 150-250 ms time window (with -100-0 ms as baseline). Score is unbounded. Larger negative values indicated a better score (i.e., larger MMN)

CONTACTS AND LOCATIONS:
Overall Officials: Arcara, Principal Investigator — IRCCS San Camillo Hospital
Locations (4):
- Italy (4):
  - IRCCS San Raffaele, Milan, MI
  - IRCCS Eugenio Medea, Pieve di Soligo, TV
  - Istituto Universitario di Studi Superiori Pavia, Pavia
  - IRCCS San Camillo Hospital, Venice

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bambini V, Agostoni G, Buonocore M, Tonini E, Bechi M, Ferri I, Sapienza J, Martini F, Cuoco F, Cocchi F, Bischetti L, Cavallaro R, Bosia M. It is time to address language disorders in schizophrenia: A RCT on the efficacy of a novel training targeting the pragmatics of communication (PragmaCom). J Commun Disord. 2022 May-Jun;97:106196. doi: 10.1016/j.jcomdis.2022.106196. Epub 2022 Feb 2. PMID 35526293